CLINICAL TRIAL: NCT02122263
Title: Transient Elastography of the Liver ( Fibroscan ) and Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Assy Nimer, Proffessor, Ziv Hospital
Other Study IDs: 0007-14-ZIV
Record Dates: First submitted 2014-03-20; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NAFLD after sleeve gastrectomy surgery

SUMMARY:
To evaluate the effect of Bariatric surgery on the extent of liver fat and liver fibrosis and on different metabolic parameters in patients undergoing sleeve gastrectomy surgery.

DETAILED DESCRIPTION:
The effect of bariatric surgery on the extent of fat and extent of liver fibrosis following sleeve gastrtrectomy is unknown. Methods : 60 obese NAFLD patients will undergo sleeve gastrectomy surgery. Measurements will be conducted at: baseline, and at 6 Month and will include: abdominal US, Fibroscan elastography , biochemical tests, anthropometric measurements, and questionnaires for demographic details, quality of life, food intake, food tolerance and habitual physical activity. Primary Outcome Measures: Liver fat quantification (controlled attenuation parameter;CAP ) and stiffness at baseline and at 6 months by fibroscan. The liver stiffness is measured by Fibroscan in a volume of approximates 1 cm wide and 4 cm long cylinder, representing 1/500 of liver tissue (100 times greater than a biopsy sample). The results of the Fibroscan will be expressed in KiloPascals (kPa). The Fibroscan XL probe reduces Fibroscan failure and facilitates reliable liver stiffness measurement in obese patients compared with the common M probe. Secondary Outcome Measures: metabolic parameters including insuline resistance, CRP, MDA, Paraoxonase, and bile acid levels. Quality of life and Food tolerance after bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-65 years old
* BMI > 40 kg/m² or BMI > 35 kg/m² with comorbidities
* Willingness to take a metformin once a day for 6 months
* Ultrasound diagnosed NAFLD patients
* Reading and speaking Hebrew

Exclusion Criteria:

* Subject with mental illness or cognitive deterioration
* Use of probiotic/antibiotic 3 mounts before surgery
* Use of other antibiotic for more than 1 week during the study
* Drug addiction
* Excessive alcohol consumption (≥ 30 g/day in men or ≥ 20 g/day in women)
* Treatment with drugs known to cause hepatic steatosis or elevation of liver enzymes (e.g. Corticosteroids, HAART, Amiodarone, high dose estrogens)
* Treatment with drugs or supplements that may improve hepatic steatosis or liver enzymes (Vitamin E, Milk thistle, ω-3 fatty acid, Ursodeoxycholic acid) 3 months prior to the initiation of the study
* Other causes of chronic liver disease ( e.g. viral hepatitis: HBV/HCV +, autoimmune hepatitis, Hemochromatosis, Wilson's disease)
* Diabetic patients who are treated with antidiabetic medications, except diabetic patients who are treated for at least 6 months exclusively with Metformin at a stable dose
* Subjects who began a new lipid reduction medications less than 6 months prior to the initiation of the study
* Subjects with chronic conditions that could interfere with our study: active cancer, organ transplant subjects, advanced kidney or liver disease, inflammatory bowel disease and other systemic inflammatory conditions
* Bariatric surgery in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 obese NAFLD patients after sleeve gastrectomy surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Transient elastography | 6 month after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nimer Assy, Prof, Principal Investigator — Ziv Medical Center
Locations (1):
- ZIv Medical Center, Safed, Israel, Israel